CLINICAL TRIAL: NCT05491291
Title: Cross-cultural and Psychometric Validation of the RESVECH 2.0 Scale for the Assessment of Chronic Wounds in the French West Indies.
Brief Title: Chronic Wound Care of Lower Limb in M@diCICAT Center at CHU de Martinique
Acronym: VALRESCIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20_RIPH23-27
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Chronic Wounds
Keywords: Chronic wounds; RESVECH 2.0; Wound assesment tool; cross-cultural validation,

STUDY DESIGN:
Intervention Model Description: The rating scale will be passed at three different times, day 1, day 15 and day 75.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chronic wound of the lower limbs (Other): Passing of the scale when the patient will come at the hospital for his routine health care visit in M@diCICAT center
  Interventions: Other: Patients with chronic wound of the lower limbs

INTERVENTIONS:
Other: Patients with chronic wound of the lower limbs — The rating scale will be passed at three different times, day 1, day 15 and day 75.

SUMMARY:
Chronic wound of lower limb. In developed countries, the prevalence of chronic wounds is linked to the ageing of the population and the increase in chronic diseases such as diabetes, obesity and cardiovascular disease. Consequence: amputations of lower limb. The prevalence of chronic wounds is also variable across the globe. In addition, chronic wounds are associated with psychosocial problems such as poor quality of life, loss of professional activity and progressive de-socialization of patients. To improve the quality of care we need in french wound assessment tools validated scientifically like the RESVECH 2.0 scale, validated in the Spanish language.

DETAILED DESCRIPTION:
The VALRESCIC study aims to perform a cross-cultural and psychometric validation of the RESVECH 2.0 scale in order to be able to use it for monitoring wounds in both hospital and primary care settings in the French West Indies.

The RESVECH 2.0 scale is a heterogeneous scale to monitor the evolution of a chronic wound. This scale was created in 2010 and consists of 6 items with response modalities ranging from 5 to 14. The interpretation of the scale parameters may differ depending on the cultural context. The RESVECH 2.0 scale has been validated in the Spanish language (in Spain and Colombia) to assess the progress towards healing of pressure ulcers and chronic wounds of the lower limbs.

For the cross-cultural evaluation we will follow Beaton's methodology, which includes: translation, synthesis, retro-translation, expert committee review and pre-testing. For the psychometric validation, the following parameters will be measured: Feasibility and acceptability, validity, reliability, and sensitivity to change.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one chronic wound of the lower limbs admitted to the M@diCICAT® healing centre.
* Patients agreeing to participate in the study
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Patients with critical ischemia of the lower limb concerned
* Patients under legal protection measures (guardianship, curatorship, safeguard of justice) and persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Cultural adaptation of the RESVECH 2.0 scale. | Before the start of recruitment
  Validation of scale RESVECH 2.0 translation in french language depending on the cultural context in French West Indies
Psychometric validation of the RESVECH 2.0 scale. | 15 days post inclusion
  Scientific validation of the french version of the scale RESVECH 2.0 in French West Indies

CONTACTS AND LOCATIONS:
Overall Officials: Maria CANO SANCHEZ, RN, Study Director — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez-Del-Rio RF. Factors Associated to the Cicatrization Success of Lower-Limb Ulcer of Venous Etiology. Invest Educ Enferm. 2018 Sep;36(3). doi: 10.17533/udea.iee.v36n3e08. PMID 31083854
- [Result] Aragon-Sanchez J, Lipsky BA, Lazaro-Martinez JL. Diagnosing diabetic foot osteomyelitis: is the combination of probe-to-bone test and plain radiography sufficient for high-risk inpatients? Diabet Med. 2011 Feb;28(2):191-4. doi: 10.1111/j.1464-5491.2010.03150.x. PMID 21219428
- See also: A Coefficient of Agreement for Nominal Scales — https://www.semanticscholar.org/paper/A-Coefficient-of-Agreement-for-Nominal-Scales-Cohen/9e463eefadbcd336c69270a299666e4104d50159
- See also: Validation des échelles d'évaluation en médecine physique et de réadaptation : comment apprécier correctement leurs qualités psychométriques — https://www.em-consulte.com/article/34264/validation-des-echelles-d-evaluation-en-medecine-p